CLINICAL TRIAL: NCT01345279
Title: Indirect Comparison of the Efficacy Between Topotecan and Other Treatments for Recurrent Carcinoma of the Cervix
Brief Title: Indirect Comparison Topotecan Cervical Carcinoma
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 114016
Record Dates: First submitted 2010-07-16; First posted 2011-05-02 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Cervical Intraepithelial Neoplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — Cisplatin; Topotecan; Paclitaxel

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- cisplatin
  Interventions: Drug: cisplatin
- cisplatin + topotecan
  Interventions: Drug: cisplatin; Drug: topotecan
- cisplatin + paclitaxel
  Interventions: Drug: cisplatin; Drug: paclitaxel

INTERVENTIONS:
Drug: cisplatin — 50 mg/m2 IV cisplatin on day 1 and then every 3 weeks for 6 courses
Drug: topotecan — topotecan 0.75 mg/m2 on days 1, 2, and 3. The regimen was repeated every 3 weeks for 6 courses
  Groups: cisplatin + topotecan
Drug: paclitaxel — 135 mg/m2 paclitaxel on day 1 and then every 3 weeks for 6 courses
  Groups: cisplatin + paclitaxel

SUMMARY:
Indirect comparisons were performed using data from GOG-0179 versus GOG-0169 to permit comparison of topotecan in combination with cisplatin versus cisplatin plus paclitaxel via the common comparator of cisplatin monotherapy. Both GOG-0179 and GOG-0169 were conducted in patients with stage IVB, recurrent or persistent carcinoma of the cervix, but there were some differences between the respective study populations. Patients with prior chemotherapy were eligible for GOG-0179 but ineligible for GOG-0169 (except when chemotherapy was used for radiation sensitisation). Fewer patients had received chemotherapy as a radiosensitiser in GOG-0169 (27%) than in GOG-0179 (~60%) and these patients were unevenly distributed between treatment arms in GOG-0169. In addition, the proportion of patients receiving cisplatin as a radiosensitiser in GOG-0169 is unknown. For these reasons, there are limitations associated with the indirect meta-analysis.

ELIGIBILITY:
Inclusion Criteria:

* randomised clinical trials, or systematic reviews and meta-analyses
* treatment with topotecan or platinum-based single and combination regimens in female patients of any race with cancer of the cervix recurrent after radiotherapy or stage IVB disease

Exclusion Criteria:

* None

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The search was designed to identify all clinical data published since the Cancer Care Ontario systematic review in 2006. The Cancer Care Ontario systematic review searched MEDLINE (1966 to February 2006), EMBASE (1980 to February 2006), the Cochrane Library (Cochrane Database of Systematic Reviews (2006 Issue 1), and Cochrane Controlled Trials Register (2006 Issue 1)), the Canadian Medical Association Infobase, and the National Guidelines Clearinghouse. The conference proceedings of the American Society of Clinical Oncology (1995-2005) and the European Society of Medical Oncology (2002-2005) were also searched. The search was completed on 18 December 2008
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2009-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Overall survival | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline